CLINICAL TRIAL: NCT04398277
Title: A Daily Coping Toolkit for Medical Personnel and First-Responders During the COVID-19 Pandemic
Brief Title: A Daily Coping Toolkit for Medical Personnel and First-Responders During COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kent State University (Other)
Responsible Party: Principal Investigator, Karin Coifman, Associate Professor, Psychological Sciences, Kent State University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-183
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Psychological Stress
Keywords: COVID-19 Pandemic
MeSH Terms: conditions — Stress, Psychological; COVID-19

STUDY DESIGN:
Intervention Model Description: All participants receive the intervention. There is a brief randomized manipulation for dosage in the first 7 days only then all participants receive the higher dose.
Who Masked: Participant, Investigator
Masking Description: Participants are randomized to dose condition without their knowledge for the first 7 days. The primary investigator is blinded to conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial Low dose (Active Comparator): Participants will receive only one daily positive emotion prompt in the first seven days of the toolkit use.
  Interventions: Behavioral: Daily Coping Toolkit
- Initial high dose (Active Comparator): Participants will receive two daily positive emotion prompts in the first seven days of use.
  Interventions: Behavioral: Daily Coping Toolkit

INTERVENTIONS:
Behavioral: Daily Coping Toolkit — 1. Emotion Labelling Activity: Participants rate 10 discrete negative and positive emotional words on a likert scale (0-4).
  2. Expressive Writing and Self Distancing Activity: Participants respond to an open-ended prompt to write about their day in an open text box in response to the prompt: "What was today like for you?" After this is completed, they are prompted that if the experience was very challenging, to revisit that experience in their mind by taking a "fly on the wall" perspective (Kross & Ayduk, 2016).
  3. Positive Emotion Generation Activity (1 v. 2 prompts) Participants are prompted to take a deep breath and then respond to 1 (or 2) of 8 possible prompts in which they can generate positive emotions. In response to each, they are asked to describe their thoughts or memories in open-ended text box.

SUMMARY:
During the current COVID-19 Pandemic, all communities are relying heavily on medical personnel and first-responders to maintain high levels of psychological and occupational functioning. However, during times of persistent high levels of stress, many individuals experience depletion in psychological resources, suffering intense distress that can make daily occupational and interpersonal functioning difficult. In order to assist with this immense challenge, this research team has developed a brief daily intervention based on decades of stress and trauma research that may help to support psychological health in individuals on the frontlines who are most essential to society. Considerable evidence supports the role of attention to and conceptualization of emotional experience in psychological resilience. This project tests a highly innovative combination of interventions targeting these processes in a brief, daily activity. The primary project aim is to investigate the Daily Coping Toolkit for medical personnel and first responders to determine efficacy over time, to test relative dosing, and to explicate the underlying therapeutic processes. The toolkit consists of 3 activities, administered one time each day, taking minutes to complete and will be administered to n=1000 personnel. Data analysis will test the impact of the toolkit on momentary affective processes and on symptoms and wellbeing over 9 months. The impact of this research will be evidence to support the further use of this novel tool to assist essential front-line personnel during this ongoing crisis helping to mitigate the psychological toll and also support occupational functioning now and in the future.

DETAILED DESCRIPTION:
During times of persistent high levels of stress, many individuals experience depletion in psychological resources, suffering intense distress that can make daily occupational and interpersonal functioning difficult. In order to assist during this exceptionally challenging crisis, this research team has developed a brief daily intervention based on decades of stress and trauma research that may help to support psychological health and coping resources in individuals on the frontlines: medical personnel and first-responders. These are individuals who are most essential to society in this difficult time. Although hospitals, fire, and police departments have existing support resources in place, they are either based on traditional models of treatment or consist of online peer-support or wellness applications. All facets of existing support/interventions have considerable utility, but it is not clear that these resources are designed to address the frequent and ongoing coping demands of this crisis across a broad swath of individuals. In particular, traditional psychotherapy models are unlikely to be successful due to very real time constraints of this population at this time. Moreover, several decades of research would argue that traditional psychotherapy is unlikely to be needed by most individuals, given prototypical patterns of adjustment across a range of aversive events, including prior pandemics (SARS: Bonanno, et al 2008). However, even resilient individuals will struggle with distress and some symptoms. Prior research has suggested that specific emotion processing patterns can support resilient outcomes over the long-term and thus frontline workers may benefit from an intervention that leverages this existing knowledge to facilitate adaptive emotion regulatory processing and elevate well-being during this crisis.

The proposed project aims to investigate a novel intervention: A Daily Coping Toolkit, administered via online application, that consists of 3 activities targeting adaptive emotional attention and expression, administered one time each day, only 4-10 minutes in duration daily. The Toolkit is both practically feasible given the demands and current burden on the target population as well as highly consistent with existing evidence. Moreover, the Toolkit is not likely to conflict with other online tools or with traditional psychotherapy and hence, can be practically applied across a broad swath of individuals in need. The primary project aim is to test the Daily Coping Toolkit on a broader population of medical personnel and first responders to determine efficacy over time, to test relative dosing, and to explicate the underlying therapeutic processes. The potential impact of this research will be evidence to support the further use of this novel tool to assist essential front-line personnel during this ongoing crisis. This may assist with mitigating the psychological toll of this crisis and also support the occupational functioning of medical personnel and first responders, thus, contributing indirectly to improved patient outcomes. Finally, knowledge gained from this research will support the further development of this tool to support individuals facing future challenging events and circumstances.

Participants: n=1000 medical personnel and first responders to test the efficacy of the Daily Coping Toolkit.

Procedure: Interested individuals will go to www.tinyurl.com/dailycopingtoolkit for additional information, including the informed consent. Once consent is provided, individuals complete a brief assessment of current symptoms, well-being and psychiatric/treatment history and then receive instructions to download the research application ExpiWell (www.expiwell.com) a secure platform that operates on ios/Android devices upon which we administer the Toolkit. Once downloaded, participants are randomized to a high versus low treatment condition and will receive daily prompts to complete the intervention. After 7 days, they complete a brief assessment of symptoms, well-being, and acceptability of the intervention and consent again for continuation in the research. Individuals can continue to use the application without consenting further if they choose and their data will not be accessible to researchers. For those that do consent, follow-up assessments occur at 2,6, and 9 months (symptoms and well-being).

Daily Coping Toolkit Intervention: Participants are prompted one time daily (with 1-2 reminders) to complete the intervention which consists of the following three parts. Randomization to high versus low condition is maintained for the first 7 days only in order to test for relative dose effects (see #3 below).

1. Emotion Labelling Activity: Participants rate 10 discrete negative and positive emotional words on a likert scale (0-4). Precise labelling of emotional experience can serve as a form of implicit emotion regulation and has been associated with healthy psychophysiological and behavioral adaptation in a range of community and clinical samples
2. Expressive Writing and Self Distancing Activity: Participants respond to an open-ended prompt to write about their day in an open text box in response to the prompt: "What was today like...?" After this is completed, they are prompted that if the experience was very challenging, to revisit that experience in their mind by taking a "fly on the wall" perspective (Kross & Ayduk, 2016; see figure for instructions). Persistent evidence has indicated that expressive writing is an effective coping tool. In addition, research has identified the ways in which specific word use can facilitate healthy emotional processing during stress. There is also significant research demonstrating that shifting perspective about negative emotional experiences can facilitate a healthier distance from it.
3. Positive Emotion Generation Activity (1 v. 2 prompts) Participants are prompted to take a deep breath and then respond to 1 (or 2) of 8 possible prompts in which they can generate positive emotions. In response to each, they are asked to describe their thoughts or memories in open-ended text box. Note: For the first 7 days, participants are randomized to either respond to one (low dose) or two (high dose) prompts so as to test the relative efficacy of the "dose". After 8 days, all participants default to the higher dose of 2 prompts. Prompts are designed to elicit gratitude, positive social experiences, amusing memories, kind acts they committed, satisfaction/pride with accomplishments, positive future focus, and love for close others. Prior research has demonstrated that positive emotions generated during highly stressful events predict resilience and improved emotion regulation and coping. Moreover, positive emotion generation has been shown broadly to predict increased psychological wellbeing.

ELIGIBILITY:
Inclusion Criteria: Active Medical Personnel or First-Responders working during the COVID-19 Pandemic -

Exclusion Criteria: NONE

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 4 | 1 week
  Patient Health Questionnaire 4 items, Kroenke, Spitzer, Williams & Lowe, 2009
Patient Health Questionnaire - 4 | 9 weeks
  Patient Health Questionnaire 4 items, Kroenke, Spitzer, Williams & Lowe, 2009
Patient Health Questionnaire - 4 | 26 weeks
  Patient Health Questionnaire 4 items, Kroenke, Spitzer, Williams & Lowe, 2009
Patient Health Questionnaire - 4 | 40 weeks
  Patient Health Questionnaire 4 items, Kroenke, Spitzer, Williams & Lowe, 2009
World Health Organization Well Being Questionnaire | 1 week
  2 items from the WHO-5: Beck 2004
World Health Organization Well Being Questionnaire | 9 weeks
  2 items from the WHO-5: Beck 2004
World Health Organization Well Being Questionnaire | 26 weeks
  2 items from the WHO-5: Beck 2004
World Health Organization Well Being Questionnaire | 40 weeks
  2 items from the WHO-5: Beck 2004
Affective Experience | 1 week
  Reported negative and positive emotions: Coifman et al, 2016
Treatment Acceptability Questionnaire | 1 week
  Adapted from Hunsley, 1992, assessed subjective experience with intervention

CONTACTS AND LOCATIONS:
Overall Officials: Doug Delahanty, PhD, Principal Investigator — Kent State University; John Gunstad, PhD, Principal Investigator — Kent State University
Locations (3):
- United States (3):
  - Akron Children's Hospital, Akron, Ohio
  - Summa Health Systems, Akron, Ohio
  - Kent State University, Kent, Ohio

IPD SHARING:
Plan to Share IPD: Yes
All data and materials will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after data collection is complete
Access Criteria: Contact the PI